CLINICAL TRIAL: NCT06830512
Title: The Safety and Efficacy Evaluation of Echocardiography-guided Percutaneous Radiofrequency Ablation for Cardiac Tumors: a Single-arm, Prospective, Single-center Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20232307-F-2
Record Dates: First submitted 2025-01-07; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-03

CONDITIONS: Heart Neoplasms
Keywords: cardiac tumors；echocardiography-guided percutaneous radiofrequency ablation; safety; efficacy
MeSH Terms: conditions — Heart Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Echocardiography-guided percutaneous radiofrequency ablation
  Interventions: Procedure: Echocardiography-guided percutaneous radiofrequency ablation for cardiac tumors

INTERVENTIONS:
Procedure: Echocardiography-guided percutaneous radiofrequency ablation for cardiac tumors — In the parasternal long-axis section, the cardiac puncture guide line was used to locate the puncture, and the best puncture path through the chest wall was selected. The coaxial biopsy needle was punctured through the guide frame, and then through the skin and subcutaneous tissue into the heart tumor tissue to take 2-10 biopsy samples, which were sent for pathological examination. The biopsy needle was extracted, and the radiofrequency electrode needle was punctured along the coaxial sheath to the planned ablation site of the heart tumor. The radiofrequency ablation device was started and the ablation treatment was performed.

SUMMARY:
The safety and efficacy evaluation of echocardiography-guided percutaneous radiofrequency ablation (Liwen prcocedure) for cardiac tumors: a single-arm, prospective, single-center clinical study.

DETAILED DESCRIPTION:
Cardiac tumor is a rare disease in clinical practice, which is divided into primary cardiac tumor and secondary cardiac tumor, of which secondary cardiac tumor is about 20 to 40 times of primary.The clinical symptoms of cardiac tumors are complex and varied, mainly related to the size and location of tumors. Tumors often lead to blood flow obstruction, arrhythmia, systemic embolism, which seriously threaten the life of patients.At present, surgical resection is the only operation treatment. However, many cardiac tumors have lost the chance of surgery because of many reasons.

Based on previous work, we found echocardiography-guided percutaneous radiofrequency ablation (Liwen procedure) to treat cardiac tumors.This is a single-arm, prospective, single-center clinical study. After signing the informed consent letter, the patients were screened to meet the enrollment conditions and were treated with Liwen procedure for cardiac tumors. Follow-up was performed at 7 days, 30 days, 3 months, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodynamic changes caused by cardiac tumors or patients with obvious clinical symptoms such as chest tightness, shortness of breath, palpitations, etc., or the risk of embolization of intracardial tumors;
2. Patients who cannot be completely excised by surgery, cannot tolerate surgery or refuse surgery;
3. The patient was informed of the nature of the clinical study and agreed to participate in all the requirements of the clinical study, signed the informed consent, and agreed to complete the follow-up and follow-up examination required.

Exclusion Criteria:

1. Previously documented persistent ventricular tachycardia or ventricular fibrillation, supraventricular tachycardia with hemodynamic disturbance, cardiac arrest, and high atrioventricular block;
2. Previous history of tumor or thromboembolism exfoliating organ embolism;
3. Combined with other heart diseases requiring surgical treatment;
4. Active infections should be treated with antibiotics;
5. Bleeding constitution and coagulation disorders, or anticoagulation, antiplatelet therapy contraindications;
6. Patients who are pregnant, breastfeeding or planning to become pregnant during the clinical study;
7. The disease will cause difficulties in the evaluation of treatment, such as mental illness, metabolic disease, etc.;
8. Patients who cannot tolerate general anesthesia;
9. Severe liver, kidney, lung, brain and other major organ failure;
10. There are no patients who are suitable for the injection path of Liwen operation;
11. Other diseases deemed unsuitable for inclusion by the researchers;
12. The researcher judged that the patients' dependence was poor and could not complete the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Effective response rate (Effective defined as ≥30% reduction in the total longest diameter of the target lesion first detected during the postoperative follow-up period and confirmed 4 weeks after surgery) | 1 year
30 days after surgery: Cardiovascular mortality | 1 year

SECONDARY OUTCOMES:
Patients benefited from 1-year overall survival (OS) and progression-free survival (PFS) | 1 year
Arrhythmia, hemodynamics, cardiac function rating (NYHA rating), and quality of life (QLQ-C30 score) were improved at 3, 6, and 12 months after surgery | 1 year
New malignant arrhythmias (persistent ventricular tachycardia or ventricular fibrillation, cardiac arrest, high atrioventricular block) | 1 year
Embolism (including stroke and systemic embolism) | 1 year
Surgery-related organ injury (including cardiac rupture) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No